CLINICAL TRIAL: NCT04102618
Title: A Window-of-opportunity Study of Pelareorep in Early Breast Cancer (AWARE-1)
Brief Title: A Window-of-opportunity Study of Pelareorep in Early Breast Cancer
Acronym: AWARE-1
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment into AWARE cohorts1-4 have concluded and the primary objective and core goals for the study were met.
Sponsor: Oncolytics Biotech (Industry)
Collaborators: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REO 027
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Breast; Breast Cancer; Primary Breast; Primary Breast Cancer; Pelareorep; Atezolizumab; Reovirus; Oncolytic virus; Letrozole; Early Breast Cancer; Triple-negative breast cancer; HR+ breast cancer; HER2+ breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — reolysin; Letrozole; atezolizumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (closed to enrollment) (Experimental): HR+/HER2-neg patients who will receive pelareorep plus letrozole
  Interventions: Biological: Pelareorep; Drug: Letrozole
- Cohort 2 (closed to enrollment) (Experimental): HR+/HER2-neg patients who will receive pelareorep plus letrozole plus atezolizumab
  Interventions: Biological: Pelareorep; Drug: Letrozole; Drug: Atezolizumab
- Cohort 3 (closed to enrollment) (Experimental): TNBC patients who will receive pelareorep plus atezolizumab
  Interventions: Biological: Pelareorep; Drug: Atezolizumab
- Cohort 4 (closed to enrollment) (Experimental): HER2+/HR+ patients who will receive pelareorep plus trastuzumab plus atezolizumab
  Interventions: Biological: Pelareorep; Drug: Atezolizumab; Drug: Trastuzumab
- Cohort 5 (closed to enrollment) (Experimental): HER2+/HR- patients who will receive pelareorep plus trastuzumab plus atezolizumab
  Interventions: Biological: Pelareorep; Drug: Atezolizumab; Drug: Trastuzumab
- Cohort 6 (Experimental): HER2+ (irrespective of HR status) (6 patients) who will receive pelareorep + trastuzumab
  Interventions: Biological: Pelareorep; Drug: Trastuzumab

INTERVENTIONS:
Biological: Pelareorep — 4.5 × 10e10 TCID50 administered intravenously on Days 1, 2, 8 & 9
  Other Names: Previously REOLYSIN®
Drug: Letrozole — Oral dose of 2.5 mg/day starting on Day 3 for 13 days
  Arms: Cohort 1 (closed to enrollment); Cohort 2 (closed to enrollment)
Drug: Atezolizumab — 1200 mg administered intravenously on Day 3
  Arms: Cohort 2 (closed to enrollment); Cohort 3 (closed to enrollment); Cohort 4 (closed to enrollment); Cohort 5 (closed to enrollment)
Drug: Trastuzumab — 8mg/kg administered intravenously or 600mg subcutaneously on Day 3
  Arms: Cohort 4 (closed to enrollment); Cohort 5 (closed to enrollment); Cohort 6

SUMMARY:
The purpose of this study is to find out if pelareorep in combination with different therapies helps to reduce the growth of breast cancer cells and increase the immune system's response to cancer. This study will also help to understand what this treatment does to the tumor. In addition, the safety of the combination treatments with pelareorep will be evaluated.

DETAILED DESCRIPTION:
This is a window of opportunity non-randomized exploratory study to evaluate the safety and anti-tumor immunogenicity of pelareorep -/+ atezolizumab in five different cohorts in women with operable early breast cancer.

After enrollment, pelareorep will be administered at 4.5 × 1010 TCID50 intravenously on days 1, 2, 8 & 9. Other therapies will be administered according to the assigned treatment cohort.

After an initial biopsy (diagnostic biopsy in most cases), a second biopsy will be performed on Day 3. Patients will continue the planned treatment until day 21(±5), when a third biopsy will be performed. This third biopsy can be the surgical specimen if patient was scheduled for primary surgery, or a core biopsy if patient will undergo neoadjuvant treatment.

Blood samples will be collected throughout the study at three time points, Day 1, Day 3, and End of Treatment.

Patients will receive treatment for 3 weeks prior to surgery or neoadjuvant therapy. Thereafter, patients will either be considered for definitive surgery or primary medical treatment (e.g. neoadjuvant chemotherapy) at the discretion of the treating physician. Surgery or biopsy prior to neoadjuvant chemotherapy should be done within 3 weeks (±5 days) from the start of the study treatment.

The end of study visit will be performed at the day of surgery. A safety follow-up, the end of study visit, will be done at 28 days (± 7 days) after the last dose of treatment received

ELIGIBILITY:
Patient Inclusion Criteria:

1. Signed written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures and assessments.
2. Female patients.
3. Age ≥18 years. In cohorts 1 and 2 (patients with HR+/HER2 negative breast cancer), only postmenopausal* patient can be included.
4. Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast, with all of the following characteristics:

   * At least 1 lesion that can be measured in at least 1 dimension with ≥ 10 mm in largest diameter measured by ultrasound and mammogram.
   * Documentation confirming the absence of distant metastasis (M0) as determined by institutional practice. Routine exams to discard metastases will be performed according to Investigator judgement but are mandatory in case of suspicion of metastatic disease.
   * Breast cancer eligible for primary surgery.
   * In the case of a multifocal tumor (defined as the presence of two or more foci of cancer within the same breast quadrant), the largest lesion must be ≥ 10 mm and designated the "target" lesion for all subsequent tumor evaluations and biopsies.
5. Patient must have biopsiable disease.
6. Histologically confirmed HER2 status and hormone receptors (ER and PgR) according to ASCO/CAP guidelines locally assessed.

   * Invasive TNBC defined as: ER and PR negative defined as IHC nuclear staining <1% AND HER2 negative.
   * HR+/HER2 negative defined as: ER and PR positive defined as IHC nuclear staining >1% AND HER 2 negatives.
   * HER2 positive defined as; IHC +++ or FISH positive.
7. ECOG Performance Status of 0 or 1.
8. Adequate organ function, as determined by the following laboratory tests, within 14 days prior to randomization:

   * Hematological

     * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
     * Platelet count ≥ 100 x 109/L
     * Hemoglobin ≥ 9 g/dL (red blood cell transfusion and/or erythropoietin allowed)
   * Renal

     o Serum creatinine ≤ 1.5 x upper limit of normal (ULN), or 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance does not need to be determined if the baseline serum creatinine is within normal limits. Creatinine clearance should be calculated per institutional standard).
   * Hepatic

     * Serum bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN
     * Aspartate aminotransferase (AST) ≤ 3 x ULN
     * Alanine aminotransferase (ALT) ≤ 3 x ULN
     * Coagulation International normalization ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN
     * Partial thromboplastin time (PTT) or activated PTT (aPTT) ≤ 1.5 x ULN
9. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (only for cohorts 3 to 5 and pre-menopausal women or non-confirmed postmenopausal* status).

    * *postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.) OR
    * have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening; OR
    * has a congenital or acquired condition that prevents childbearing.

Patient Exclusion Criteria

1. Inoperable locally advanced or inflammatory (i.e., inoperable Stage III) breast cancer.
2. Metastatic (Stage IV) breast cancer.
3. Bilateral invasive breast cancer.
4. Multicentric breast cancer, defined as the presence of two or more foci of cancer in different quadrants of the same breast.
5. Prior therapy for breast cancer.
6. Prior therapy with an anti- PD-1, anti- PD-L1, anti-PD-L2, anti-CD137 antibody, or anti-CTLA-4 antibody compound, Pelareorep or any other oncolytic viruses.
7. Prior therapy with tumor vaccine
8. History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease, or active autoimmune disease or syndrome that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs) except vitiligo or resolved childhood asthma/atopy or evidence of clinically significant immunosuppression. Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Treated or untreated hyperthyroidism. Uncontrolled hypothyroidism (patients with controlled and asymptomatic hypothyroidism can be included)
10. Received any vaccine, including against SARS-COV-2 (COVID-19), <14 days prior to the first day of study treatment. Inactivated vaccines (including against COVID-19 or seasonal influenza) are permitted after surgery.
11. History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other malignancies with an expected curative outcome.
12. Evidence of clinically significant immunosuppression such as the following:

    * diagnosis of immunodeficiency
    * concurrent opportunistic infection
    * receiving systemic immunosuppressive therapy (> 2 weeks) or within 7 days prior to the first dose of study treatment, including oral steroid doses > 10 mg/day of prednisone or equivalent. Subjects that require intermittent use of bronchodilators or local steroid injection will not be excluded from the study.
13. Cardiopulmonary dysfunction as defined by:

    * Uncontrolled hypertension (systolic >150 mm Hg and/or diastolic > 100 mm Hg) despite optimal medical management.
    * Inadequately controlled angina or serious cardiac arrhythmia not controlled by adequate medication.
    * History of symptomatic congestive heart failure (CHF): Grade ≥ 3 per NCI CTCAE version 4.03 or Class ≥ II New York Health Association (NYHA criteria).
    * Myocardial infarction within 6 months prior to randomization.
    * Current dyspnea at rest due to complications of advanced malignancy, or other disease requiring continuous oxygen therapy
14. Current severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary or metabolic disease; wound healing disorders; ulcers; bone fractures).
15. Major surgical procedure or significant traumatic injury within approximately 28 days prior to enrollment or anticipation of the need for major surgery during the course of study treatment.
16. Concurrent, serious, uncontrolled infections or current known infection with HIV or active hepatitis B and/or hepatitis C.
17. Assessment by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
18. Known history of active Bacillus tuberculosis.
19. History of significant co-morbidities that, in the judgment of the Investigator, may interfere with the conduction of the study, the evaluation of response, or with informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
To evaluate if pelareorep in combination with different therapies increases the value of the CelTIL score in women with operable early breast cancer. CelTIL is a combined IHC-based score based on tumor cellularity and stromal TILs. | The CelTIL score will be measured from on-treatment tumor biopsies collected at baseline (pre-treatment), day 3, and at time of surgery (day ~21 ± 5 days).
  CelTIL score is a metric for quantifying broad changes to the tumor microenvironment and is calculated by the following equation:
  CelTIL score = -0.8 × tumor cellularity (in percent) + 1.3 × TILs (in percent). The minimum and maximum unscaled CelTIL scores will be -80 and 130. This unscaled CelTIL score will then be scaled to reflect the reported values ranging from 0 to 100 points where an increase in CelTIL scores represent favorable changes to the tumor microenvironment.

SECONDARY OUTCOMES:
To evaluate if pelareorep in combination with different therapies increases the value of the CelTIL score in women with HR+/HER2-negative breast cancer. | The CelTIL score will be measured from on-treatment tumor biopsies collected at baseline (pre-treatment), day 3, and at time of surgery (day ~21 ± 5 days).
To evaluate if pelareorep in combination with different therapies increases the value of the CelTIL score in women with HER2-positive breast cancer. | The CelTIL score will be measured from on-treatment tumor biopsies collected at baseline (pre-treatment), day 3, and at time of surgery (day ~21 ± 5 days).
To identify biological changes, as defined by gene expression between posttreatment and pretreatment samples following pelareorep in combination with different therapies. | throughout
To describe the safety profile of the combination therapies | throughout

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - ICO Badalona, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Quirón Dexeus, Barcelona
  - Hospital Moisés Broggi, Esplugues de Llobregat
  - Hospital Fuenlabrada, Madrid
  - Hospital La Paz, Madrid
  - Hospital Puerta de Hierro de Majadahonda, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Clínico Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza